CLINICAL TRIAL: NCT05283434
Title: Arnica and the Management of Pain in Acute Musculoskeletal Extremity Injuries
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Principal Investigator, Manu Madhok, Physician, Children's Hospitals and Clinics of Minnesota
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1812-139
Record Dates: First submitted 2022-03-07; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Pain, Muscle; Pain, Acute
Keywords: Homeopathy; Pain Management; Musculoskeletal Extremity Injuries; Swelling
MeSH Terms: conditions — Myalgia; Acute Pain; Agnosia | interventions — Arnicae flos extract

STUDY DESIGN:
Intervention Model Description: Double-Blind Clinical Trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double-Blind Clinical Trial- Placebo Group (Placebo Comparator): Patients will be assigned to the placebo (e.g., unmedicated sugar pill) or experimental group (e.g., Arnica 1M pellets) via a randomization chart from that only the research pharmacist will have access to. Subjects assigned to the placebo group will take the recommended doses of sugar pellets (i.e., 2 pills to be taken every 4 waking hours over a 24 hours period), and will track their pain scores, swelling measurements, sleep rate, ibuprofen doses, adverse reactions, further ED visits, and the number of days/activities the patient has missed for 3 days following their enrollment in the study.
  Interventions: Drug: Placebo
- Double-Blind Clinical Trial- Experimental Group (Experimental)
  Interventions: Drug: Arnica

INTERVENTIONS:
Drug: Arnica — Patients will be assigned to the placebo (e.g., unmedicated sugar pill) or experimental group (e.g., Arnica 1M pellets) via a randomization chart from that only the research pharmacist will have access to. Subjects assigned to the experimental group will take the recommended doses of Arnica 1M coated sugar pellets (i.e., 2 pills to be taken every 4 waking hours over a 24 hours period), and will track their pain scores, swelling measurements, sleep rate, ibuprofen doses, adverse reactions, further ED visits, and the number of days/activities the patient has missed for 3 days following their enrollment in the study.
  Arms: Double-Blind Clinical Trial- Experimental Group
Drug: Placebo — Sugar pill placebo
  Arms: Double-Blind Clinical Trial- Placebo Group

SUMMARY:
In the Emergency Department, there is no standard of care for pain medication distribution for children with an acute musculoskeletal injury when there is no fracture present. Currently, ibuprofen is a favorable choice for the treatment, but studies have shown concern for delayed healing activity associated with NSAIDs like Ibuprofen. Homeopathic Arnica Montana is a well-established complimentary medicine and may provide a good alternative for managing acute pain from musculoskeletal injuries, especially in children, given the palatability and rarity of side effects. This study aims to compare usual care vs. usual care plus Arnica 1M* (oral) or the placebo for management of pain in acute musculoskeletal extremity injuries without fracture by utilizing a double-blind clinical trial design. The primary outcome is to determine if subjects use less ibuprofen when given Arnica 1M.

ELIGIBILITY:
Inclusion Criteria:

* Patient presents to the Emergency Department with an acute, soft tissue ankle or forearm injury
* ED Provider orders an X-ray for evaluation of injury
* Patient's initial pain score is of a 4 or higher
* Patient has noticeable swelling at the site of the injury

Exclusion Criteria:

* Patient is diagnosed with a fracture
* Patient has an allergy to ibuprofen
* Patient is already on a NSAID, acetaminophen, anticoagulant or oral corticosteroid therapy for chronic pain treatment (a NSAID given in triage or use for the current injury is allowed)
* Use of other concurrent complementary medicine therapy, e.g. massage, acupuncture, physical therapy
* Patient has been treated for this injury in the past
* Patient has a bleeding/bruising disorder
* Patient is pregnant or is lactating
* Patient has a liver or kidney disease, malignancy, infection, immunodeficiency or metabolic syndrome
* Patient is allergic to the Asteraceae family of plants (arnica, ragweed, chrysanthemum, marigold, or daisy are the most common)
* Patient is nonverbal, and thus unable to give a pain score
* Patient does not have a working telephone (required for follow-up call)
* Family requires foreign language interpreter during their ED visit

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 324 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Ibuprofen Dose | Initial Emergency Department Visit to three full days after discharge
  Amount of Ibuprofen the patient consumed during the three full days after discharge

SECONDARY OUTCOMES:
Swelling | Initial Emergency Department Visit to three full days after discharge
  Swelling Measurement (cm)
Pain Score | Initial Emergency Department Visit to three full days after discharge
  Patient's Pain Score on a 1-10 scale where 1 is the lowest
Arnica Dosage | Within the first 24 hours of discharge
  The amount of Arnica doses (e.g., 2 pills) that were consumed; ranging from 1 to 4.

OTHER OUTCOMES:
Routine Change | Three full days after discharge
  The number of days the family's usual routine has been changed or disrupted following discharge
Days of School/Work family members missed | Three full days after discharge
  The number of days of school and/or work days the patient's family missed after discharge
Days of School/Activities that a patient has missed | Three full days after discharge
  The number of days of school and/or activities the patient missed after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Manu Madhok, MD, MPH, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (2):
- United States (2):
  - Children's Minnesota, Minneapolis, Minnesota
  - Children's Minnesota, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
There is no plan in place to make individual participant data available to other researchers.

REFERENCES:
- [Background] Thompson EA, Bishop JL, Northstone K. The use of homeopathic products in childhood: data generated over 8.5 years from the Avon Longitudinal Study of Parents and Children (ALSPAC). J Altern Complement Med. 2010 Jan;16(1):69-79. doi: 10.1089/acm.2009.0007. PMID 20105063
- [Background] Oberbaum M, Schreiber R, Rosenthal C, Itzchaki M. Homeopathic treatment in emergency medicine: a case series. Homeopathy. 2003 Jan;92(1):44-7. doi: 10.1054/homp.2002.0071. PMID 12587994
- [Background] Arnica. 2024 Oct 15. Drugs and Lactation Database (LactMed(R)) [Internet]. Bethesda (MD): National Institute of Child Health and Human Development; 2006-. Available from http://www.ncbi.nlm.nih.gov/books/NBK501828/ PMID 30000888
- [Background] Mawardi H, Ghazalh S, Shehatah A, Abdelwahid A, Aljohani A, Felemban O, Almazrooa S, Elbadawi L, Shawky H. Systemic Use of Arnica Montana for the Reduction of Postsurgical Sequels following Extraction of Impacted Mandibular 3rd Molars: A Pilot Study. Evid Based Complement Alternat Med. 2020 Dec 12;2020:6725175. doi: 10.1155/2020/6725175. eCollection 2020. PMID 33381206
- [Background] Iannitti T, Morales-Medina JC, Bellavite P, Rottigni V, Palmieri B. Effectiveness and Safety of Arnica montana in Post-Surgical Setting, Pain and Inflammation. Am J Ther. 2016 Jan-Feb;23(1):e184-97. doi: 10.1097/MJT.0000000000000036. PMID 25171757
- [Background] Paris A, Gonnet N, Chaussard C, Belon P, Rocourt F, Saragaglia D, Cracowski JL. Effect of homeopathy on analgesic intake following knee ligament reconstruction: a phase III monocentre randomized placebo controlled study. Br J Clin Pharmacol. 2008 Feb;65(2):180-7. doi: 10.1111/j.1365-2125.2007.03008.x. PMID 18251757
- [Background] Karow JH, Abt HP, Frohling M, Ackermann H. Efficacy of Arnica montana D4 for healing of wounds after Hallux valgus surgery compared to diclofenac. J Altern Complement Med. 2008 Jan-Feb;14(1):17-25. doi: 10.1089/acm.2007.0560. PMID 18199022
- [Background] Robertson A, Suryanarayanan R, Banerjee A. Homeopathic Arnica montana for post-tonsillectomy analgesia: a randomised placebo control trial. Homeopathy. 2007 Jan;96(1):17-21. doi: 10.1016/j.homp.2006.10.005. PMID 17227743
- [Background] Brinkhaus B, Wilkens JM, Ludtke R, Hunger J, Witt CM, Willich SN. Homeopathic arnica therapy in patients receiving knee surgery: results of three randomised double-blind trials. Complement Ther Med. 2006 Dec;14(4):237-46. doi: 10.1016/j.ctim.2006.04.004. Epub 2006 Oct 13. PMID 17105693

DOCUMENTS (1):
  • Study Protocol (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT05283434/Prot_000.pdf